CLINICAL TRIAL: NCT05156450
Title: Phase Ib/II Clinical Study of TQB3616 Capsules in Combination With Abiraterone Acetate Plus Prednisone in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: TQB3616 Capsules Combined With Abiraterone Acetate Plus Prednisone in Metastatic Castration-Resistant Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Hao Zeng, Professor of Department of Urology, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMPA 2018L02262/2018L02263
Record Dates: First submitted 2021-11-19; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Prostatic Neoplasms, Castration-Resistant; Drug Therapy, Combination
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Extension (Experimental): At the recommended phase II dose of TQB3616 combined with abiraterone acetate (1000 mg, q.d.) plus prednisone (5 mg, b.i.d.), 20-40 patients are planned to be enrolled to evaluate the efficacy and safety of the combination therapy.
  Metastatic and genomic tests based on tissue biopsy samples (primary or metastatic) and blood samples will be performed before treatment and after disease progression.
  Interventions: Drug: TQB3616 Capsules Combined With Abiraterone Acetate Plus Prednisone

INTERVENTIONS:
Drug: TQB3616 Capsules Combined With Abiraterone Acetate Plus Prednisone — Treatment with TQB3616 in combination with abiraterone acetate plus prednisone in patients with metastatic castration-resistant prostate cancer.

SUMMARY:
This is a phase Ib/II clinical study of TQB3616 capsules in combination with abiraterone acetate plus prednisone in patients with metastatic castration-resistant prostate cancer, to determine the dose for further clinical studies and to evaluate the safety and efficacy of this combined therapy.

DETAILED DESCRIPTION:
TQB3616 is an inhibitor of Cyclin-dependent kinases 4 and 6 (CDK4/6), which reduces intracellular protein phosphorylation levels, prevents cells from entering synthesis (S) phase from first gap (G1) phase, and inhibits cell proliferation to combat tumors. TQB3616 has superior inhibitory activity to Palbociclib and Abemaciclib against CDK4/6 kinase and may benefit metastatic castration-resistant prostate cancer (mCRPC) patients through a complementary mechanism of action when combined with abiraterone acetate plus prednisone. Therefore, the investigators intend to perform this phase Ib/II clinical study of TQB3616 capsules in combination with abiraterone acetate plus prednisone in patients with mCRPC.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients ≥ 18 years old and ≤ 80 years old (based on the date of signed informed consent); willing and able to provide written informed consent and good compliance.
2. Histologically or cytologically confirmed prostatic adenocarcinoma. Patients with small cell or large cell neuroendocrine carcinoma, prostatic uroepithelial carcinoma, basal cell carcinoma, sarcomatoid carcinoma, carcinoid carcinoma and ductal adenocarcinoma are excluded.
3. Imaging (e.g. bone scan and CT/MRI) confirmed metastatic disease.
4. Serum testosterone level ≤ 1.73 nmol/L (50 ng/dL) at the screening visit. Patients who did not undergo bilateral orchiectomy required continued treatment with androgen deprivation therapy (ADT) [gonadotropin-releasing hormone analogue (LHRHa, agonist/antagonist)] throughout the study period.
5. Disease progression during/post consecutive ADT, as determined at the time of study inclusion, defined as meeting one or more of the following criteria:

   1. At least two consecutive elevated PSA values separated by at least 1 week, and if elevated PSA is determined to be the only evidence of progression, the last result must be at least 1.0 ng/mL. Patients receiving anti-androgen therapy must have experienced PSA progression after discontinuation (≥4 weeks since last flutamide administration or ≥6 weeks since last bicalutamide or nilumet).
   2. Disease progression as assessed by RECIST 1.1, regardless of the presence of PSA progression.
   3. Skeletal disease progression as assessed by PCWG3, i.e. ≥ 2 new lesions found on bone scan and re-evaluated at least 8 weeks later with ≥ 2 new lesions other than the last evaluated new bone lesions, regardless of the presence of PSA progression.
6. Patients must have discontinued all prior cancer therapy (except ADT and bone loss prophylaxis) and have recovered to ≤ Grade 1 or baseline (according to the Common Terminology Criteria for Adverse Events version 5.0 [CTCAE v 5.0]) from all acute toxic effects of prior therapy or surgery prior to the first dose, except alopecia and peripheral neuropathy, and the washout period since the last previous systemic or radiation therapy is as follows:

   1. At least 4 weeks must have elapsed from the use of 5-alpha reductase inhibitors (e.g., dutasteride, finasteride), estrogens, and cyproterone to enrollment.
   2. At least 4 weeks must have elapsed from the use of chemotherapy (i.e., docetaxel for metastatic hormone sensitive prostate cancer) to enrollment.
   3. At least 4 weeks must have elapsed between major surgery or radiation therapy and enrollment.
7. Normal organ function (including blood routine, blood biochemistry, urine routine, coagulation function, thyroid function, cardiac function assessment, etc.).
8. Eastern Cooperative Oncology Group (ECOG) physical status (PS) of 0 to 1. Expected survival ≥ 6 months.
9. Willingness to comply with study procedures. Patients of childbearing potential must agree to use an effective method of contraception and avoid sperm donation for the duration of the study and for at least 3 months after the last study treatment dose.

Exclusion Criteria:

Those who present any of the following criteria will not be enrolled in this trial.

1. Tumor disease and medical history.

   1. Subjects with brain metastases with symptoms or symptom control for less than 1 month, unless signs and/or symptoms of central nervous system (CNS) involvement are present, screening for CNS metastases is not required at baseline.
   2. Have presented within 3 years or have a current concurrent other malignancy. The following two conditions are eligible for enrollment: other malignancies treated with a single procedure to achieve 5 consecutive years of disease free generation (DFS); cured carcinoma in situ of the cervix, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)]; for patients with carcinoma in situ of any origin and for patients with previous malignancies currently in remission are eligible to participate in this study if, in the judgment of the investigator, the likelihood of recurrence is considered very low, and the investigator will approve these patients prior to enrollment.
   3. Those whose imaging (CT or MRI) shows that the tumor has invaded the vital vascular perimeter or who, in the judgment of the investigator, are at high risk of fatal hemorrhage due to tumor invasion of vital vessels during the follow-up study.
   4. the presence of severe bone damage caused by tumor bone metastases; or pathological fractures and spinal cord compression at important sites that have occurred within the last 6 months or are expected to be likely to occur in the near future as judged by the investigator.
   5. uncontrolled pleural effusion, pericardial effusion or ascites that still requires repeated drainage (in the judgment of the investigator).
2. Prior antitumor or combination drug therapy.

   1. Use of botanicals (e.g., saw palmetto) that may lower PSA levels within 4 weeks prior to the first dose.
   2. Prior antineoplastic therapy less than 4 weeks from the first dose, including surgery, chemotherapy, palliative radiotherapy for non-target lesions, hormonal therapy (including first-generation AR antagonists [e.g., flutamide, bicalutamide, nilumide], 5α-reductase inhibitors [e.g., finasteride], estrogens, and cyproterone), adjuvant therapy with targeted agents, biologic therapy, cytokine immunotherapy, clinical trial drug therapy, etc.
   3. previous oral targeted drugs with less than 5 drug half-lives from the first dose (calculated from the end time of the last treatment)
   4. Prior antitumor therapy-related toxicity not recovered to Common Terminology Criteria for Adverse Events (CTCAE) ≤ grade 1, except for alopecia.
   5. Previous treatment with cytochrome P450 family 17 (CYP17) inhibitors (including agents such as TAK-700, TOK-001 and ketoconazole), with no restrictions for patients previously treated with abiraterone.
   6. Prior treatment with Abemaciclib or Palbociclib and any other CDK4/6 inhibitors.
   7. Patients treated with drugs known to be potent inhibitors of cytochrome P450 3A4 (CYP3A4) or potent or moderately potent inducers and unable to discontinue these drugs or switch to a different drug at least 5 half-lives prior to initiation of study drug therapy.
3. Co-morbidities and medical history.

   1. Liver abnormalities.

      * Decompensated cirrhosis (Child-Pugh liver function rating of B or C).
      * Active or chronic hepatitis [Hepatitis B reference: Hepatitis B surface antigen (HBsAg) positive with Hepatitis B virus (HBV) DNA test value exceeding the upper limit of normal; Hepatitis C reference: Hepatitis C virus (HCV) antibody positive with HCV viral titer test value exceeding the upper limit of normal]; Hepatitis B surface antigen-positive or core antibody-positive eligible enrolled subjects, hepatitis C subjects, who require continuous antiviral therapy to prevent viral activation.
      * Patients with ascites or bleeding disorders secondary to hepatic insufficiency.
   2. Renal abnormalities.

      * Renal failure requiring hemodialysis or peritoneal dialysis.
      * Previous history of nephrotic syndrome.
   3. Cardiovascular abnormalities.

      * History of epilepsy, or history of seizures, impaired consciousness or transient ischemic attack within the last 12 months, or history of unexplained coma.
      * Class II to IV heart failure as defined by the New York Heart Association classification, or heart ejection fraction < 50% at baseline. Second degree or greater heart block, myocardial infarction or arterial thrombosis event within the last 6 months, unstable arrhythmia or unstable angina.
      * Cerebrovascular accident, cerebral infarction, etc. within 6 months.
      * Presence of hypertension not controlled by medication (at least 2 measurements of ≥ 150 mmHg systolic and ≥ 100 mmHg diastolic); for patients with a history of hypertension, participation in this study is allowed if blood pressure is adequately controlled by antihypertensive therapy.
      * Previous or current cardiac valvulitis, endocarditis.
      * syncope of cardiovascular origin, pathological ventricular arrhythmias (including but not limited to ventricular tachycardia and ventricular fibrillation), or sudden cardiac death.
   4. Gastrointestinal abnormalities.

      * Inability to take oral medications (e.g., inability to swallow, chronic diarrhea, and intestinal obstruction).
      * History of malabsorption syndrome or other conditions that would interfere with gastrointestinal absorption.
      * Treatment for active peptic ulcer or ulcerative lower gastrointestinal inflammation within the past 6 months.
      * Persistent chronic diarrhea of grade 2 or greater despite maximal medical therapy.
      * Investigator-determined conditions that may cause other conditions that may cause gastrointestinal bleeding or perforation, as determined by the investigator.
   5. History of immunodeficiency.

      * Known human immunodeficiency virus (HIV) infection.
      * Other acquired, congenital immunodeficiency disorders.
      * Preparation for or previous organ transplantation, or hematopoietic stem cell transplantation within 60 days prior to first dose, or with significant host transplantation response.
      * Need for immunosuppressive, or systemic, or absorbable local hormone therapy for immunosuppression purposes and Patients requiring immunosuppressive, or systemic, or absorbable topical hormone therapy for immunosuppression and requiring continued use for 7 days prior to the first dose (except for glucocorticoids at doses <10 mg prednisone daily or other isotonic hormones)
   6. Bleeding risk.

      * Patients with bleeding (hemoptysis), coagulopathy or on warfarin, aspirin and other anti-platelet coagulation drugs (except aspirin ≤100 mg/d prophylaxis).
      * Patients with any physical signs or history of bleeding, regardless of severity.
      * Any CTCAE ≥ grade 3 bleeding or bleeding event within 4 weeks prior to the first dose.
   7. Patient has an active systemic infection (e.g., bacterial infection requiring intravenous antibiotic therapy at the time of initiation of study treatment, fungal infection, or detectable viral infection requiring systemic therapy) or viral load (e.g., known human immunodeficiency virus positivity or known active hepatitis B or C [e.g., hepatitis B surface antigen positivity]. Screening for this is not required to determine eligibility for enrollment.
   8. History of idiopathic pulmonary fibrosis, history of histoplasmosis (e.g., occlusive fine bronchitis), history of drug-induced pneumonia, history of idiopathic pneumonia, or evidence of active pneumonia on screening-period CT scan of the chest.
   9. Allergy or previous history of severe allergy; or known hypersensitivity to study drug excipient components.
   10. Previous history of definite neurological or psychiatric disorder.
   11. Combination of a serious or poorly controlled disease that the investigator determines may be at greater risk for entry into this study [e.g., type 1 or type 2 diabetes mellitus not controlled by medication, thyroid disease].
   12. History of pituitary or adrenal gland dysfunction.
   13. Major surgical treatment, incisional biopsy or significant traumatic injury within 28 days prior to the start of study treatment.
   14. Long-term untreated wounds or fractures.
   15. History of substance abuse or drug use.
4. Participation in another drug clinical trial within the previous 30 days or current enrollment in a clinical study involving an experimental product, or enrollment in any other type of medical study judged to be scientifically or medically incompatible with this study. Have participated in any clinical trial in which treatment assignment remains blinded, and if the patient is currently enrolled in a clinical trial involving an unapproved use of a medical device, concurrence of the investigator and the Center is required to determine Eligibility for enrollment.
5. Recent live vaccination (within 4 weeks prior to the first dose). Receipt of inactivated vaccine is permitted.
6. Insufficient estimated patient compliance to participate in this clinical study.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
12-month radiographic progression-free survival (rPFS) rate | 12 months
  Percentage of subjects with radiographic progression-free survival of 12 months or more

SECONDARY OUTCOMES:
rPFS | 2 years
  Radiographic progression-free survival: Refers to the time between the start of enrollment and the onset of disease imaging progression or recurrence or death from all causes, whichever occurs first. Imaging-confirmed disease progression includes: soft tissue and lymph node disease progression as evaluated by Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1), and bone metastases progression as evaluated by the Prostate Cancer Working Group 3 (PCWG3) .
6-month rPFS rate | 6 months
  Percentage of subjects with radiographic progression-free survival of 6 months.
Prostate specific antigen (PSA) response rate | 2 years
  The percentage of subjects whose PSA decrease by more than 50% of the baseline value and maintain for more than 4 weeks.
Time to PSA progression | 2 years
  The time from the first dose to the confirmation of PSA progression. The PCWG3 standard defines PSA progression as: For subjects with a ≥50% decrease in PSA at 12 weeks of treatment, a 25% increase in PSA above the nadir and an absolute increase of ≥2 ng/mL compared to the nadir, and confirmed by a second PSA test ≥3 weeks later; for subjects with a non-responsive PSA at 12 weeks of treatment, a 25% increase in PSA above baseline and an absolute increase of ≥2 ng/mL compared to the baseline value, and confirmed by a second PSA test ≥3 weeks later.
Objective response rate (ORR) | 2 years
  Objective response rate: The percentage of subjects in complete response (CR) or partial response (PR) as determined by the investigator according to RECIST 1.1.
Overall survival (OS) | 2 years
  Overall survival: The time between the start of enrollment and death from all causes.
Clinical benefit rate (CBR) | 2 years
  Clinical benefit rate: The best overall outcome (BOR) was the proportion of stable disease (SD) subjects with CR, PR and duration ≥24 weeks as rated by RECIST 1. 1 criteria.
Duration of response (DOR) | 2 years
  Duration of response: For subjects whose best remission was CR or PR, this is defined as the time between the date of first documented tumor remission and the date of first documented disease progression or death from any cause, whichever occur first.

OTHER OUTCOMES:
Biomarkers related to efficacy, mechanism of action, safety, and/or pathogenesis, such as cell cycle pathway-related genes | 2 years
  Biomarker consistency in tumor tissue samples versus blood samples and correlation between biomarkers with efficacy will be analyzed. Biological samples will be collected during the screening period and out of the group, and tested by second-generation sequencing technology. The selected genes are all reported to be related to cell cycle pathways, such as RB1, CDK4/6, CDKN2A (p16 INK4a), CDKN2B (p15 INK4b), CDKN2C (p18 INK4c) and CDKN2D (p19 INK4d), and genes related to AR, TP53, DNA repair pathway, PI3K/AKT signaling pathway, WNT signaling pathway and MAPK signaling pathway, etc., which have been reported to be relevant to prostate cancer treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zeng, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Background] Center MM, Jemal A, Lortet-Tieulent J, Ward E, Ferlay J, Brawley O, Bray F. International variation in prostate cancer incidence and mortality rates. Eur Urol. 2012 Jun;61(6):1079-92. doi: 10.1016/j.eururo.2012.02.054. Epub 2012 Mar 8. PMID 22424666
- [Background] Knudsen ES, Witkiewicz AK. The Strange Case of CDK4/6 Inhibitors: Mechanisms, Resistance, and Combination Strategies. Trends Cancer. 2017 Jan;3(1):39-55. doi: 10.1016/j.trecan.2016.11.006. PMID 28303264
- [Background] Kase AM, Copland Iii JA, Tan W. Novel Therapeutic Strategies for CDK4/6 Inhibitors in Metastatic Castrate-Resistant Prostate Cancer. Onco Targets Ther. 2020 Oct 15;13:10499-10513. doi: 10.2147/OTT.S266085. eCollection 2020. PMID 33116629
- [Background] First CDK 4/6 Inhibitor Heads to Market. Cancer Discov. 2015 Apr;5(4):339-40. doi: 10.1158/2159-8290.CD-NB2015-028. Epub 2015 Feb 23. PMID 25711280
- [Background] Comstock CE, Augello MA, Goodwin JF, de Leeuw R, Schiewer MJ, Ostrander WF Jr, Burkhart RA, McClendon AK, McCue PA, Trabulsi EJ, Lallas CD, Gomella LG, Centenera MM, Brody JR, Butler LM, Tilley WD, Knudsen KE. Targeting cell cycle and hormone receptor pathways in cancer. Oncogene. 2013 Nov 28;32(48):5481-91. doi: 10.1038/onc.2013.83. Epub 2013 May 27. PMID 23708653
- [Background] Frank S, Nelson P, Vasioukhin V. Recent advances in prostate cancer research: large-scale genomic analyses reveal novel driver mutations and DNA repair defects. F1000Res. 2018 Aug 2;7:F1000 Faculty Rev-1173. doi: 10.12688/f1000research.14499.1. eCollection 2018. PMID 30135717